CLINICAL TRIAL: NCT01626573
Title: A Double- Blind, Placebo Controlled Study Exploring the Safety, Tolerability, and Efficacy of a 28 Day Course Followed by an Additional 56 Day Course of Itacitinib in Subjects With Active Rheumatoid Arthritis
Brief Title: A Study Exploring the Safety, Tolerability, and Efficacy of a 28 Day Course Followed by an Additional 56 Day Course of Itacitinib in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39110-201
Record Dates: First submitted 2012-05-03; First posted 2012-06-22 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; Active
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — itacitinib; INCB039110

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- Itacitinib 400 mg twice a day (Experimental): Itacitinib 400 mg twice a day
  Interventions: Drug: Itacitinib
- Itacitinib 400 mg placebo twice a day (Placebo Comparator): Itacitinib 400 mg placebo twice a day
  Interventions: Drug: Itacitinib Placebo
- Itacitinib 100 mg twice a day (Experimental): This dose group will be studied twice during the study.
  Interventions: Drug: Itacitinib
- Itacitinib 100 mg placebo twice a day (Placebo Comparator): This dose group will be studied twice during the study.
  Interventions: Drug: Itacitinib Placebo
- Itacitinib 100mg once a day (Experimental): Itacitinib 100mg once a day
  Interventions: Drug: Itacitinib
- Itacitinib 100 mg placebo once a day (Placebo Comparator): Itacitinib 100 mg placebo once a day
  Interventions: Drug: Itacitinib Placebo
- Itacitinib 200 mg twice a day (Experimental): Itacitinib 200 mg twice a day
  Interventions: Drug: Itacitinib
- Itacitinib 200 mg placebo twice a day (Placebo Comparator): Itacitinib 200 mg placebo twice a day
  Interventions: Drug: Itacitinib Placebo
- Itacitinib 300 mg once a day (Experimental): Itacitinib 300 mg once a day
  Interventions: Drug: Itacitinib
- Itacitinib 300 mg placebo once a day (Placebo Comparator): Itacitinib 300 mg placebo once a day
  Interventions: Drug: Itacitinib Placebo
- Itacitinib 600 mg once a day (Experimental): Itacitinib 600 mg once a day
  Interventions: Drug: Itacitinib
- Itacitinib 600 mg placebo once a day (Placebo Comparator): Itacitinib 600 mg placebo once a day
  Interventions: Drug: Itacitinib Placebo

INTERVENTIONS:
Drug: Itacitinib
  Other Names: INCB039110
  Arms: Itacitinib 100 mg twice a day; Itacitinib 100mg once a day; Itacitinib 200 mg twice a day; Itacitinib 300 mg once a day; Itacitinib 400 mg twice a day; Itacitinib 600 mg once a day
Drug: Itacitinib Placebo
  Arms: Itacitinib 100 mg placebo once a day; Itacitinib 100 mg placebo twice a day; Itacitinib 200 mg placebo twice a day; Itacitinib 300 mg placebo once a day; Itacitinib 400 mg placebo twice a day; Itacitinib 600 mg placebo once a day

SUMMARY:
This is a study evaluating a 28-day course followed by a 56-day course of itacitinib in patients with active rheumatoid arthritis (RA). The study will evaluate safety and efficacy parameters of itacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with active RA aged 18 to 75 years of age and meet tender and swollen joint assessment expectations defined in the study protocol.
* c-Reactive protein (CRP) or erythrocyte sedimentation rate (ESR) laboratory values meet minimal study protocol expectations.

Exclusion Criteria:

* Females who are pregnant or breastfeeding.
* Men and women who cannot comply with requirements to avoid fathering a child or becoming pregnant, respectively.
* Subjects treated with a biologic agent within 12 weeks prior to first dose of study drug. (12 months in the case of rituximab.)
* Subjects with a history or currently suspected inflammatory disease other than RA.
* Subjects with a history of hematological disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of itacitinib as assessed by the changes in frequency and severity of adverse events, ECGs, vital signs, physical examinations, and clinical laboratory evaluations. | Approximately four months.
Preliminary efficacy as assessed by the percentage of patients achieving ACR20 improvement from baseline on the day 28 and day 84 visits. | Approximately 84 days.

SECONDARY OUTCOMES:
Preliminary Pharmacokinetic (PK) collections. | Following 15 days of therapy.
  Plasma concentrations of itacitinib will be used to estimate peak plasma concentration (Cmax) and area under the plasma concentration-time curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Sandor, MD, Study Director — Incyte Corporation
Locations (18):
- United States (17):
  - Palm Desert, California
  - Pasadena, California
  - Lake Mary, Florida
  - Ocala, Florida
  - Palm Harbor, Florida
  - Tampa, Florida
  - Tavares, Florida
  - Lexington, Kentucky
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Raleigh, North Carolina
  - Middleburg Heights, Ohio
  - Duncansville, Pennsylvania
  - Florence, South Carolina
  - Austin, Texas
  - Katy, Texas
  - Spokane, Washington
- Carolina, Puerto Rico